CLINICAL TRIAL: NCT00473109
Title: Chronic Hemodialysis Without Systemic Heparinization : a Randomized Study
Acronym: HDSH
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Responsible Party: Christophe AUCAN, Department Clinical Rechearch of Developpement
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: P050311; CRC05032
Record Dates: First submitted 2007-05-11; First posted 2007-05-14 (Estimated); Last update posted 2009-05-25 (Estimated); Status verified 2007-05

CONDITIONS: Contra-Indication to the Use of Low Molecular Weight Heparin
Keywords: Hemodialysis; Heparin; Clotting
MeSH Terms: conditions — Thrombosis | interventions — Dialysis

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Dialysis without systemic heparinization (Experimental): Dialysis without systemic heparinization
  Interventions: Procedure: Dialysis without systemic heparinization

INTERVENTIONS:
Procedure: Dialysis without systemic heparinization — Dialysis without systemic heparinization

SUMMARY:
Conventional hemodialysis requires transient systemic anticoagulation to prevent blot clotting after contact with the extracorporeal circuit. However, low molecular weight heparin (LMWH) or unfractioned heparin are contra-indicated in dialysis patients at risk for hemorrhagic complications. In this setting, several procedures theoretically allow dialysis without systemic heparinization, but randomized studies to compare them are lacking. The gold standard is the use of iterative rises of the extra corporeal circuit with isotonic saline (" rises "). Two emerging procedures are increasingly used : continuous pre-dilution of the arterial line (" pre-dilution ") and the use of a specific dialysis membrane (NEPHRAL 400 ST) coated with heparin immediately before use (" heparin adsorption ").

DETAILED DESCRIPTION:
Conventional hemodialysis requires transient systemic anticoagulation to prevent blot clotting after contact with the extracorporeal circuit. However, low molecular weight heparin (LMWH) or unfractioned heparin are contra-indicated in dialysis patients at risk for hemorrhagic complications. In this setting, several procedures theoretically allow dialysis without systemic heparinization, but randomized studies to compare them are lacking. The gold standard is the use of iterative rises of the extra corporeal circuit with isotonic saline (" rises "). Two emerging procedures are increasingly used : continuous pre-dilution of the arterial line (" pre-dilution ") and the use of a specific dialysis membrane (NEPHRAL 400 ST) coated with heparin immediately before use (" heparin adsorption ").

We propose a monocentric prospective randomized open study to compare " rises ", " pre-dilution " and " heparin adsorption " in chronic hemodialysis patients with contra-indication to the use of LMWH. Main criteria will be extra-corporeal circuit clotting, with dialysis efficiency and tolerance as secondary criteria. Comparison will be made on grounds of " n-of-1 " trial, i.e. series of randomized cross-over tests in individuals. We have planned to include 75 patients in this study, with 1050 LMWH-free dialysis sessions.

We hope to demonstrate chat by comparison wit rises, pre-dilution and heparin absorption techniques reduce the rate of extra-corporeal circuit by 30 and 50% respectively. We also hope to show that heparin adsorption (i) better preserves membrane integrity throughout the dialysis session, resulting in enhanced dialysis efficiency ; (ii) avoids extra fluid infusion and ultrafiltration, resulting in better dry weigh achievement and better clinical tolerance.

ELIGIBILITY:
Inclusion Criteria:

* Chronic hemodialysis patient
* Low molecular weight heparin contra indicated for at least 3 consecutive hemodialysis sessions.

Exclusion Criteria:

* Acute renal failure
* Access flow < 250 ml/mn)
* Per dialytic Blood transfusion or parenteral nutritional support
* Systolic BP < 80 mm Hg
* Hemoglobin > 13 g/dl

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 75 (Actual)
Dates: Start 2007-05; Primary Completion 2009-03 (Actual); Study Completion 2009-05 (Actual)

PRIMARY OUTCOMES:
Need for stopping the meeting for coagulation of the circuit of dialysis: -either complete coagulation of the circuit | during dialises
or coagulation partial of the circuit (a clot is noted in the lines or the trap with bubbles | during dialeses
-or increase in the venous pressure (statement) of the circuit of more than 50 that is to say increase in the venous pressure (statement) of the circuit of more than 50 % beyond its initial value | during the dialeses

SECONDARY OUTCOMES:
Loss of effectiveness of dialysis? dialysance of urea during the meeting (online measurement carried out by the generator of dialysis) | during the dialeses
Loss of effectiveness of dialysis overloads hydro-sodic persistent (weight of the patient at the end of the meeting: + 500 grams compared to the basic weight) | during the dialeses
Tolerance of the meeting of dialysis clinical side effects (cephalgias, cramps, arterial hypotension | during the dialeses
Tolerance of the meeting of dialysis hemorrhagic accidents to at the time the 48 hours following the meeting of dialysis | 48 hours following the meeting of dialysis

CONTACTS AND LOCATIONS:
Overall Officials: Dominique JOLY, MD,PhD, Principal Investigator — Assistance Publique Hopitaux de Paris
Locations (1):
- Chu de Necker, Paris, France

REFERENCES:
- [Derived] Natale P, Palmer SC, Ruospo M, Longmuir H, Dodds B, Prasad R, Batt TJ, Jose MD, Strippoli GF. Anticoagulation for people receiving long-term haemodialysis. Cochrane Database Syst Rev. 2024 Jan 8;1(1):CD011858. doi: 10.1002/14651858.CD011858.pub2. PMID 38189593
- [Derived] Guery B, Alberti C, Servais A, Harrami E, Bererhi L, Zins B, Touam M, Joly D. Hemodialysis without systemic anticoagulation: a prospective randomized trial to evaluate 3 strategies in patients at risk of bleeding. PLoS One. 2014 May 13;9(5):e97187. doi: 10.1371/journal.pone.0097187. eCollection 2014. PMID 24825343